CLINICAL TRIAL: NCT01452659
Title: A Phase II, Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled Study of the Efficacy and Safety of TAK-385 10, 20, and 40 mg (p.o.) in the Treatment of Uterine Fibroids
Brief Title: Efficacy and Safety of TAK-385 in the Treatment of Uterine Fibroids
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-385/CCT-001; U1111-1123-6815 (Registry Identifier: WHO); JapicCTI-111590 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2011-08-31; First posted 2011-10-17 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: Uterine Fibroids
Keywords: Drug Therapy
MeSH Terms: conditions — Leiomyoma | interventions — relugolix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- TAK-385 10 mg QD (Experimental)
  Interventions: Drug: TAK-385
- TAK-385 20 mg QD (Experimental)
  Interventions: Drug: TAK-385
- TAK-385 40 mg QD (Experimental)
  Interventions: Drug: TAK-385
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAK-385 — TAK-385 10 mg, tablets, orally, once daily for up to 12 weeks.
  Arms: TAK-385 10 mg QD
Drug: TAK-385 — TAK-385 20 mg, tablets, orally, once daily for up to 12 weeks.
  Arms: TAK-385 20 mg QD
Drug: TAK-385 — TAK-385 40 mg, tablets, orally, once daily for up to 12 weeks.
  Arms: TAK-385 40 mg QD
Drug: Placebo — TAK-385 placebo-matching tablets, orally, once daily for up to 12 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy and safety of TAK-385, once daily (QD), for 12 weeks in women with uterine fibroids.

DETAILED DESCRIPTION:
This study is a Phase II, multicenter, randomized, double-blind, parallel-group, placebo-controlled for evaluation of the efficacy and safety of TAK-385 10, 20, and 40 mg (p.o.) following once daily administration for 12 weeks in women with uterine fibroids.

ELIGIBILITY:
Inclusion Criteria:

1. The participant has been diagnosed with uterine fibroids and has never received surgical treatment for the myoma.
2. The participant is a premenopausal woman.
3. The participant has one or more measurable noncalcified myomas confirmed by transvaginal sonography.
4. The participant has experienced regular menstrual cycles
5. The participant is diagnosed as menorrhagia

Exclusion Criteria:

1. Participants with a screening Hb <8 g/dL
2. Participants with a previous or current history of blood disorders
3. Participants with a known history of severe hypersensitivity or severe allergy to sanitary goods
4. Participants with lower abdominal pain due to irritable bowel syndrome or severe interstitial cystitis
5. Participants with a previous or current history of thyroid dysfunction
6. Participants with a previous or current history of pelvic inflammatory disease
7. Participants with a positive PAP smear test result
8. Participants with a history of panhysterectomy or bilateral oophorectomy
9. Participants judged by investigator to have marked abnormal uterine bleeding or anovulatory bleeding
10. Participants with a previous or current history of a malignant tumor
11. Participants who have been treated with any of the following drugs: anticoagulant drug, antiplatelet drug, tranexamic acid, selective estrogen receptor modulator (SERM), activated vitamin D, other vitamin D, calcitonin, ipriflavone, steroid hormone, vitamin K, teriparatide, or denosumab
12. Participants who have been treated with any of the following drugs: oral contraceptive and sex hormone preparation, gonadotropin-releasing hormone (GnRH) analogue, dienogest, danazol, or aromatase inhibitor
13. Participants who have been treated with a bisphosphonate preparation
14. Participants with a previous or current history of severe hypersensitivity or severe allergy to drugs
15. Participants with non-diagnosable abnormal genital bleeding
16. Participants with a previous or current history of osteoporosis, bone mass loss, or other metabolic bone diseases
17. Participants with clinically significant cardiovascular disease or uncontrollable hypertension
18. Participants judged by investigator to be inappropriate to participate in this study based on the 12-lead electrocardiogram (ECG) findings
19. Participants with active liver disease or jaundice, or with alanine aminotransferase (ALT), aspartate aminotransferase (AST), or total bilirubin > 1.5 times the upper limit of normal (ULN)

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2011-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Decrease in menstrual blood loss | Week 12 (one menstrual cycle)
  Blood loss will be assessed using the Pictorial Blood Loss Assessment Chart (PBAC).

SECONDARY OUTCOMES:
Decrease in menstrual blood loss | Up to Week 6
  Blood loss will be assessed using PBAC
Decrease in menstrual blood loss | Up to Week 12.
  Blood loss will be assessed using PBAC
Amenorrhea | Week 12 (one menstrual cycle).
  Amenorrhea will be assessed using PBAC
Amenorrhea | Up to Week 6.
  Amenorrhea will be assessed using PBAC
Amenorrhea | Up to Week 12.
  Amenorrhea will be assessed using PBAC
Change in menstrual blood loss | Week 12 (one menstrual cycle)
  Change in menstrual blood loss measured by PBAC
Myoma Volume | Up to Week 12.
Uterine Volume | Up to Week 12.
Hemoglobin Concentration in Blood | Up to Week 12.
Pain Symptom | Up to Week 12.
  Measured by Numerical Rating Scale.
Other Clinical Symptoms | Up to Week 12.
  Assessed by clinical laboratory tests
Quality of Life (QOL) Score | Up to Week 12.
  QOL will be assessed using Uterine Fibroid Symptom and Quality of Life (UFS-QOL)
Bone Mineral Density | Up to Week 12.
  Measured by Dual-energy X-ray absorptiometry (DXA)
Treatment-emergent Adverse Events | Up to Week 16.
  Treatment-emergent adverse events are defined as any unfavorable and unintended sign, symptom or disease temporally associated with the use of a medicinal product reported from first dose of study drug through the last visit (Week 16)
Vital Signs | Up to Week 12.
  Vital signs will include body temperature, sitting blood pressure, and pulse (bpm).
Body Weight | Up to Week 12.
Electrocardiograms
  Up to Week 12.
Laboratory Values | Up to Week 12
Serum NTx | Up to Week 12
  NTx is one of the biochemical bone metabolism markers
Serum BAP | Up to Week 12
  BAP is one of the biochemical bone metabolism markers

CONTACTS AND LOCATIONS:
Overall Officials: Senior Director, Study Director — Takeda
Locations (27):
- Japan (27):
  - Chiba, Chiba
  - Itchihara-shi, Chiba
  - Matsuno-shi, Chiba
  - Matsuyama, Ehime
  - Nihama-shi, Ehime
  - Fukui-shi, Fukui
  - Fukuoka, Fukuoka
  - Iizuka-shi, Fukuoka
  - Yanagigawa-shi, Fukuoka
  - Mebashi-shi, Gunma
  - Ebetsu-shi, Hokkaido
  - Sapporo, Hokkaido
  - Amagasaki-shi, Hyōgo
  - Kobe, Hyōgo
  - Kamakura-shi, Kanagawa
  - Yokohama, Kanagawa
  - Ōita, Oita Prefecture
  - Ibaraki-shi, Osaka
  - Osaka, Osaka
  - Sakai-shi, Osaka
  - Tondabayashi-shi, Osaka
  - Chuo-ku, Tokyo
  - Itabashi-ku, Tokyo
  - Setagaya-ku, Tokyo
  - Shinagawa-ku, Tokyo
  - Suginami-ku, Tokyo
  - Toyama, Toyama

REFERENCES:
- [Derived] Hoshiai H, Seki Y, Kusumoto T, Kudou K, Tanimoto M. Relugolix for oral treatment of uterine leiomyomas: a dose-finding, randomized, controlled trial. BMC Womens Health. 2021 Oct 28;21(1):375. doi: 10.1186/s12905-021-01475-2. PMID 34711224